CLINICAL TRIAL: NCT05344404
Title: NR-SAFE: a Safety Study Investigating Treatment With High-dose Nicotinamide Riboside (NR) in Parkinson's Disease
Brief Title: NR-SAFE: Safety of High-dose Nicotinamide Riboside (NR) in Parkinson's Disease
Acronym: NR-SAFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/379218
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; NAD metabolism; Mitochondria; Nicotinamide Riboside
MeSH Terms: conditions — Parkinson Disease | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized double-blinded study. 20 participants randomized in 1:1 ratio to either vitamin supplementation or placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both participants and all investigators are blinded during the trial and during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nicotinamide Riboside (Experimental): Nicotinamide riboside 3000mg daily for the duration of the trial (4 weeks). Administered in tablet form in doses of 1500mg twice daily.
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo (Placebo Comparator): Placebo, no active ingredients. Administered in tablet form twice daily for the duration of the trial (4 weeks).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — 3000mg total daily. Administered in capsule form in doses of 1500mg twice daily for the duration of the trial (4 weeks).
  Other Names: Niagen; NR
  Arms: Nicotinamide Riboside
Dietary Supplement: Placebo — Placebo drug. Administered in tablet form twice daily for the duration of the trial (4 weeks).
  Arms: Placebo

SUMMARY:
NR-SAFE is a double-blinded randomized safety study aiming to determine the safety and tolerability of nicotinamide riboside (NR) at a daily dose of 3000mg, in individuals with Parkinson's disease (PD).

The investigators recently reported the results of the NADPARK study (ClinicalTrials.gov: NCT03816020), a phase I randomized, double-blinded trial, assessing the tolerability, cerebral bioavailability and molecular effects of NR therapy, 1000mg daily, in PD. The NADPARK study showed that NR 1000mg daily was well tolerated and led to a significant, but variable, increase in cerebral NAD levels (measured by 31phosphorous magnetic resonance spectroscopy, 31P-MRS) and related metabolites in the cerebrospinal fluid (CSF). NR recipients showing increased brain NAD levels exhibited altered cerebral metabolism, measured by 18fluoro-deoxyglucose positron emission tomography (FDG-PET), and this was associated with mild clinical improvement. The results of the NADPARK trial nominate NR as a potential neuroprotective therapy for PD, warranting further investigation in larger trials.

It is plausible that any beneficial effects of NR in PD may be dose-dependent and more pronounced at higher doses. NR doses of up to 2000mg daily have been tested in healthy humans with no signs of toxicity. However, the safety and tolerability of even higher doses is untested. To enable clinical studies assessing higher doses, the investigators will assess the safety and tolerability of an oral dose of 3000 mg NR daily.

NR-SAFE will recruit 20 participants with PD and randomize them 1:1 to either NR 3000mg daily or placebo for a total duration of 4 weeks.

DETAILED DESCRIPTION:
NR-SAFE is a double-blinded randomized safety study aiming to determine the safety and tolerability of nicotinamide riboside (NR) at a daily dose of 3000mg, in individuals with Parkinson's disease (PD). Individuals with PD (n = 20) will be recruited starting April 2022. Participants will be randomized 1:1 to either NR 3000mg daily (1500mg x 2) or placebo per os for a total duration of 4 week. Both the participants and the investigators will be blinded.

Primary Objective:

To determine the safety of oral NR 3000mg daily for a period of 4 weeks in individuals with Parkinson's disease (PD). Safety is defined as the absence of clinically significant NR-associated moderate or severe adverse events (AE).

Secondary Objectives:

1. Determine whether oral NR 3000 mg daily is associated with mild AE.
2. Assess the effects of oral NR 3000 mg daily on the NAD metabolome in blood and urine.
3. Assess the effects of oral NR 3000 mg daily on clinical severity of PD, measured by UPDRS.

Exploratory Objectives:

1. Assess the effects of oral NR 3000 mg daily on serum homocysteine levels.
2. Assess the effects of oral NR 3000 mg daily on fasting blood glucose and serum insulin levels.

Procedures:

After the baseline visit, participants will be reassessed in person on day 5, 7, 14, 21 and 28 by one of the neurologists involved in the study and by telephone on day 3 and 35 by the study nurse. Participants will be screened for any adverse effects on each of these consultations. Drawing of blood samples will be performed on baseline and day 3, 5, 7, 14, 21 and 28. Clinical examination and measurement of vital parameters will be performed on baseline and on day 7, 14, 21 and 28.

Primary Outcome:

Incidence of treatment-associated moderate and severe AEs.

Secondary Outcomes:

1. Between-group difference in treatment associated mild AEs.
2. Between-group difference in changes of the NAD metabolome in blood and urine, measured by mass spectrometry (LC-MS/MS Q-Exactive HF).
3. Between-group difference in change of clinical severity of PD, measured by UPDRS.

Exploratory Outcomes:

1. Between-group difference in the change of serum homocysteine levels.
2. Between-group difference in the change of fasting blood glucose and serum insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 35 years and lower than 100 years at time of enrollment.
* Clinical diagnosis of idiopathic PD according to the MDS criteria.
* Hoehn and Yahr score < 4 at enrolment.

Exclusion Criteria:

* Dementia or other neurodegenerative disorder at baseline visit.
* Any psychiatric disorder that would interfere with compliance in the study.
* Any severe somatic illness that would make the individual unable to comply and participate in the study.
* Use of high dose vitamin B3 supplementation within 30 days of enrollment.
* Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-29 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-associated moderate and severe adverse events (AEs). | 4 weeks.
  The incidence of treatment-associated moderate and severe adverse events (AEs) will be assessed.

SECONDARY OUTCOMES:
Incidence of treatment-associated mild adverse events (AEs). | 4 weeks.
  The incidence of treatment-associated mild adverse events (AEs) will be assessed.
Between-group (NR vs placebo) difference in changes of the NAD metabolome in blood and urine, measured by mass spectrometry (LC-MS/MS Q-Exactive HF) | 4 weeks.
  The concentration of NAD metabolites, such as NAD, NAAD, NAM, meNAM, etc, will be determined in blood (snap-frozen EDTA) and urin using liquid chromatography mass spectrometry (LC-MS/MS Q-Exactive HF). The change in the concentration of NAD metabolites in the NR and placebo group, as well as the between-group (NR vs placebo) difference in the change of the concentration of NAD metabolites will be assessed.
Between-group (NR vs placebo) difference in change of clinical severity of PD, measured by UPDRS. | 4 weeks.
  The change in total UPDRS in the NR and placebo group, as well as the between-group (NR vs placebo) difference in the change of total UPDRS will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berven H, Kverneng S, Sheard E, Sognen M, Af Geijerstam SA, Haugarvoll K, Skeie GO, Dolle C, Tzoulis C. NR-SAFE: a randomized, double-blind safety trial of high dose nicotinamide riboside in Parkinson's disease. Nat Commun. 2023 Nov 28;14(1):7793. doi: 10.1038/s41467-023-43514-6. PMID 38016950